CLINICAL TRIAL: NCT00170261
Title: Early Loop-Recorder in Suspected Arrhythmogenic Syncope
Brief Title: ELIAS: Early Loop-Recorder in Suspected Arrhythmogenic Syncope
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CEN_G_CA_4
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2018-04

CONDITIONS: Syncope
Keywords: Syncope of uncertain etiology; Repeated presyncopes
MeSH Terms: conditions — Syncope

INTERVENTIONS:
Device: Use of an Implantable Loop Recorder

SUMMARY:
This is a prospective, controlled, opened randomized study to evaluate the cost benefit of a primary implantation of a loop recorder versus the conventional diagnostic cascade for syncope most likely due to cardiac arrhythmia.

ELIGIBILITY:
Inclusion Criteria:

* Two or more episodes of syncope (most likely due to cardiac arrhythmia) of uncertain etiology within the last 12 months or more than one syncope and two presyncopes

Exclusion Criteria:

* Indication for the implantation of a pacemaker
* Indication for the implantation of an implantable cardioverter defibrillator
* Cardiac diseases which need intervention (KHK, aortic stenosis, mitral stenosis, left ventricular [LV] outflow stenosis, decompensated heart failure)
* Contraindication for a diagnostic procedure requested by the study protocol
* Enrollment in another study
* Circumstances or comorbidities which do not allow enrollment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2002-04; Primary Completion 2005-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Cost of diagnostics per patient until final cardiac diagnosis has been made

SECONDARY OUTCOMES:
Cost of diagnostics until final diagnosis has been made
Rate of correct cardiac diagnoses
Comparison of time needed to make a diagnosis
Comparison of pre-syncopes and syncopes occuring in both groups after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: H.-C- Ehlers, MD, Principal Investigator — Vivantes Klinikum am Urban
Locations (3):
- Germany (3):
  - Vivantes Klinikum am Urban, Berlin
  - Humbold Klinikum, Berlin
  - Universitätsklinikum Hamburg Eppendorf, Hamburg